CLINICAL TRIAL: NCT00834262
Title: A Multi Centre, Open Label, Non-Randomized, Non Interventional, Observational Study on the Safety and Efficacy of Biphasic Insulin Aspart (NovoMix® 30, NovoMix® 50 and NovoMix® 70 or Combinations) in Type 2 Diabetes Mellitus Patients
Brief Title: Observational Study on Safety and Efficacy of Biphasic Insulin Aspart in Type 2 Diabetes Patients
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-3669
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: biphasic insulin aspart 30; Drug: biphasic insulin aspart 50; Drug: biphasic insulin aspart 70

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
  Other Names: NovoMix® 30
Drug: biphasic insulin aspart 50 — Dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
Drug: biphasic insulin aspart 70 — Dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation

SUMMARY:
This study is conducted in Asia. The aim of this observational study is to evaluate the safety profile and clinical effectiveness of using various pre-mixes of Biphasic Insulin Aspart under routine clinical practice conditions in Israel in Type 2 Diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with type 2 diabetes who has HbA1c greater than 7% on insulin with or without OAD and who needs intensification of treatment with either NovoMix® 30 or NovoMix® 50 or NovoMix® 70 or combinations, will be eligible

Exclusion Criteria:

* Subjects with a hypersensitivity to biphasic insulin aspart or to any of the excipients. Particular attention should be paid to the drug interactions that are listed within the product local label.
* Women who are pregnant, breast feeding or have the intention of becoming pregnant within the next 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with type 2 diabetes who has HbA1c greater than 7% on insulin with or without OAD and who needs intensification of treatment with either NovoMix® 30, NovoMix® 50 or NovoMix® 70 or combinations, will be eligible A nonrandomized sample of approximately 325 subjects with Type 2 diabetes mellitus will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 339 (Actual)
Dates: Start 2009-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Number of all hypoglycaemic episodes | during 13 weeks of treatment

SECONDARY OUTCOMES:
Number of adverse drug reactions | during 13 weeks of treatment
Number of adverse events | during 13 weeks of treatment
Number of all major hypoglycaemic (daytime and nocturnal) episodes | during 13 weeks of treatment
Number of all minor and symptomatic (daytime and nocturnal) hypoglycaemic episodes | during 13 weeks of treatment
Number of major hypoglycaemic episodes related to omission of a meal after injection | during 13 weeks of treatment
Number of major hypoglycaemic episodes related to physical exercise of at least 30 min duration | during 13 weeks of treatment
Weight (BMI) change | at the end of the study after 13 weeks of treatment
HbA1c change | at the end of the study after 13 weeks of treatment
Percentage of patients reaching the target of HbA1c of 7.0% or less | at the end of the study after 13 weeks of treatment
Variability in fasting blood glucose values and average (mean) fasting blood glucose level | at the end of the study after 13 weeks of treatment
Average post-breakfast (2h), post-lunch (2h), post-dinner (2h) blood glucose level | at the end of the study after 13 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Kfar Saba, Israel

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com